CLINICAL TRIAL: NCT00438256
Title: Phase I/II of Neoadjuvant Accelerated Short Course Radiation Therapy With Proton Beam and Capecitabine for Resectable Pancreatic Cancer
Brief Title: Neoadjuvant Accelerated Short Course Radiation Therapy With Proton Beam and Capecitabine for Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-248
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-12

CONDITIONS: Pancreatic Cancer
Keywords: accelerated short course; proton beam radiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Proton Therapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 10 Radiation Sessions over 2 weeks
  Interventions: Procedure: Proton Beam Radiation; Drug: Capecitabine
- Group 2 (Experimental): 5 Radiation sessions: 3 in week 1 and 2 in week 2
  Interventions: Procedure: Proton Beam Radiation; Drug: Capecitabine
- Group 3 (Experimental): 5 Radiation sessions: 4 in week 1 and 1 in week 2
  Interventions: Procedure: Proton Beam Radiation; Drug: Capecitabine
- Group 4 (Experimental): 5 Radiation Sessions in one week
  Interventions: Procedure: Proton Beam Radiation; Drug: Capecitabine

INTERVENTIONS:
Procedure: Proton Beam Radiation — Given over different schedules and duration
Drug: Capecitabine — Given orally starting on day one of radiation therapy for 2 weeks

SUMMARY:
A standard treatment for pancreatic cancer is radiation therapy plus chemotherapy after surgery. Radiation therapy and chemotherapy are commonly given for up to six weeks. Previous research has suggested that giving the radiation and chemotherapy for a shorter amount of time (accelerated schedule) before surgery may be better tolerated. In this research study, different schedules of proton radiation therapy will be used. Each schedule will give about the same total dose of radiation. However, the total dose will be spread out over different time periods and different numbers of sessions. The purpose is to find the shortest schedule of radiation therapy that can be given without unacceptable side effects. Proton beam radiation is being used because of its unique ability to deposit its energy directly in the tumor, resulting in less radiation to normal tissue. A new type of PET scan is also being studied to see if it can help predict the response to pre-surgery treatment.

DETAILED DESCRIPTION:
* Not everyone who participates in this research study will receive the same schedule of radiation therapy. The schedule of radiation therapy will depend on the number of participants enrolled on the study and how well they have tolerated their radiation schedule. All patients will receive proton beam therapy.
* Here are the proposed schedules of radiation therapy. If at any point too many subjects experience too many unacceptable side effects, no subject will be enrolled to the next level. Dose Level 1: 10 radiation sessions given Monday-Friday for two weeks. Dose Level 2: 5 radiation sessions given Monday, Wednesday and Friday in Week 1 and Tuesday and Thursday in Week 2. Dose Level 3: 5 radiation sessions given Monday, Tuesday, Thursday and Friday in Week 1 and Monday in Week 2. Dose Level 4: 5 Radiation sessions given Monday through Friday in Week 1.
* In Dose Levels 2, 3 and 4, there are fewer radiation sessions, but the radiation dose given at each session is slightly higher than the dose given in each of the 10 sessions of Dose Level 1.
* Capecitabine will be given orally (pill form) starting on the first day of radiation therapy and will be taken for the two weeks that the participant receives radiation therapy.
* On days 1, 8 and 15 of each study cycle, the participant will be seen at the clinic for: physical examination, questions about side effects; and routine blood tests.
* After the last day of study treatment there will be up to a six-week rest period before surgery is performed.
* About three to six weeks after the participant has finished study treatment, the following procedures will be done: CT or MRI, physical examination; questions about side effects and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic of histologic proof of pancreatic ductal carcinoma
* No evidence of metastatic disease
* 18 years of age or older
* ECOG Performance Status of 0 or 1 - Lab values as outlined in the protocol

Exclusion Criteria:

* Tumors in the body or tail of the pancreas
* Hepatic or peritoneal metastases detected by imaging or laparoscopy prior to chemoradiation
* Serious concomitant systemic disorders incompatible with the study, such as significant cardiac or pulmonary morbidity, ongoing infection as manifested by fever
* Pregnant or lactating women
* Life expectancy of < 3 months
* Serious, uncontrolled, concurrent infection (s)
* Prior chemotherapy or radiation for treatment of the patient's pancreatic tumor
* Clinically significant cardiac disease or myocardial infarction within the last 12 months
* Other serious uncontrolled medical condition that the investigator feels might compromise study participation
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing uncontrolled coagulopathy
* Any prior fluoropyrimidine therapy
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to a 5-fluorouracil or known DPD deficiency
* Participation in any investigational drug study within 4 weeks preceding the start of the study
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery
* Patients on cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Hong TS, Ryan DP, Borger DR, Blaszkowsky LS, Yeap BY, Ancukiewicz M, Deshpande V, Shinagare S, Wo JY, Boucher Y, Wadlow RC, Kwak EL, Allen JN, Clark JW, Zhu AX, Ferrone CR, Mamon HJ, Adams J, Winrich B, Grillo T, Jain RK, DeLaney TF, Fernandez-del Castillo C, Duda DG. A phase 1/2 and biomarker study of preoperative short course chemoradiation with proton beam therapy and capecitabine followed by early surgery for resectable pancreatic ductal adenocarcinoma. Int J Radiat Oncol Biol Phys. 2014 Jul 15;89(4):830-8. doi: 10.1016/j.ijrobp.2014.03.034. Epub 2014 May 24. PMID 24867540

RESULTS

PARTICIPANT FLOW:
Groups:
- Proton Beam Radiation/ Capecitabine Dose Level 1: Procedure/Surgery:
  Proton Beam Radiation: Given over 10 Radiation Sessions over 2 weeks
  Drug:
  Capecitabine: Given orally starting on day one of radiation therapy for 2 weeks
- Proton Beam Radiation/ Capecitabine Dose Level 2: Procedure/Surgery:
  Proton Beam Radiation: Given over 5 Radiation sessions: 3 in week 1 and 2 in week 2
  Drug:
  Capecitabine: Given orally starting on day one of radiation therapy for 2 weeks
- Proton Beam Radiation/ Capecitabine Dose Level 3: Procedure/Surgery:
  Proton Beam Radiation: Given over 5 Radiation sessions: 4 in week 1 and 1 in week 2
  Drug:
  Capecitabine: Given orally starting on day one of radiation therapy for 2 weeks
- Proton Beam Radiation/ Capecitabine Dose Level 4: Procedure/Surgery:
  Proton Beam Radiation: Given over 5 Radiation Sessions in one week
  Drug:
  Capecitabine: Given orally starting on day one of radiation therapy for 2 weeks
Period: Overall Study
Arm/Group | Proton Beam Radiation/ Capecitabine Dose Level 1 | Proton Beam Radiation/ Capecitabine Dose Level 2 | Proton Beam Radiation/ Capecitabine Dose Level 3 | Proton Beam Radiation/ Capecitabine Dose Level 4
Started | 3 | 3 | 3 | 41
Surgical Resection | 1 | 2 | 2 | 34
Completed | 1 | 2 | 2 | 32
Not Completed | 2 | 1 | 1 | 9
Not completed — Ineligible for Resection | 2 | 1 | 1 | 7
Not completed — Excluded final Diagnosis | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Phase 1 radiation schedule escalation arms were combined with the phase II dose arm to highlight overall trends of the regimen
Groups:
- Proton Beam Radiation/ Capecitabine: Procedure/Surgery:
  Proton Beam Radiation: Given over different schedules and duration
  Drug:
  Capecitabine: Given orally starting on day one of radiation therapy for 2 weeks
Arm/Group | Proton Beam Radiation/ Capecitabine
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 65 [49 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
CA19-9 level at baseline [Median (Full Range); unit: units per milliliter] — Carbohydrate antigen (CA) 19-9 is an antigen released by pancreatic cancer cells.
  units per milliliter | 136.5 [1 to 15151]
Tumor size on CT [Median (Full Range); unit: Centimeters] | 2.9 [1.1 to 4.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities in the 5 Radiation Sessions in One Week Arm
Description: The number of participants that experienced a dose limiting toxicity in the arm where radiation was administered over 5 consecutive for a total dose of 25 Gray Equivalents (GyE) (Group 4). Participants were monitored for potential Dose Limiting Toxicities (DLT) for three weeks after the start of radiation. DLTs included:
  1. Any grade 3 non-hematologic or hematologic toxicity requiring a greater than 7 day interruption in therapy (excluding alopecia and nausea/vomiting not controlled by optimal supportive care or
  2. Any grade 4 non-hematologic toxicity or
  3. Any grade 4 neutropenia or thrombocytopenia as defined by Common Terminology Criteria for Adverse Events (CTCAE v3.0)
Time Frame: 3 Weeks
Population: The participants treated with radiation therapy at the 5 fractions over 5 consecutive days
Measure: Count of Participants; unit: Participants
Groups:
- Proton Beam Radiation/ Capecitabine: Procedure/Surgery:
  Proton Beam Radiation: 5 fractions over 5 consecutive days for a total of 25 Gray Equivalents (GyE)
  Drug:
  Capecitabine: Given orally starting on day one of radiation therapy for 2 weeks
Arm/Group | Proton Beam Radiation/ Capecitabine
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Number of Participants With Grade 3 or Greater Toxicity in Phase II
Description: Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE 3). The regimen was considered to be tolerated if less than 20% of participants experienced a grade 3 or greater toxicity.
Time Frame: 30 days after the end of treatment, up to approximately 6 months total
Population: Participants in the Phase II portion of the trial
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: Proton Beam Radiation/ Capecitabine: Procedure/Surgery:
  Proton Beam Radiation: 5 fractions over 5 consecutive days for a total of 25 Gray Equivalents (GyE)
  Drug:
  Capecitabine: Given orally starting on day one of radiation therapy for 2 weeks
Arm/Group | Phase II: Proton Beam Radiation/ Capecitabine
Number analyzed (Participants) | 35
Participants | 2

3. Secondary Outcome: Number of Participants With a Pathological Complete Response
Description: All patients that received surgery underwent a full pathological review of their pancreaticoduodenectomy specimen according to the American Joint Committee on Cancer (AJCC) Staging Classification, 6th. Initial gross evaluation and identification of resection margins was performed jointly by the surgeon and the pathologist. Pathological complete response will be defined as the absence of any viable tumor cells within the pathologic specimen.
Time Frame: at the time of surgery (28-42 days after start of treatment)
Population: The eligible participants who underwent surgical resection. The phase I arms and Phase II group were combined together for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Beam Radiation/ Capecitabine
Number analyzed (Participants) | 37
Participants | 0

4. Secondary Outcome: Median Progression Free Survival
Description: The median amount of time from the start of treatment until death or disease progression, whichever occurs first.
  Progressive Disease (PD): A 20% or greater increase in the sum of Longest Diameter (LD) of all target lesions, taking as reference the smallest sum LD recorded since baseline.
Time Frame: from the start of treatment until death or progression, median duration of 10.4 months
Population: Two participants were excluded from the analysis because of ineligible final diagnoses (cholangiocarcinoma and autoimmune pancreatitis)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Proton Beam Radiation/ Capecitabine
Number analyzed (Participants) | 48
Months | 10.4 [7.5 to 17.1]

5. Secondary Outcome: Number of Participants With Surgical Morbidity
Description: Number of participants with pancreatic or any other anastomotic leakage within 30 days of surgery
Time Frame: 30 days post surgery (surgery was 28-42 days after the start of treatment)
Population: The eligible participants who underwent surgical resections. The phase I arms and Phase II group were combined together for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Beam Radiation/ Capecitabine
Number analyzed (Participants) | 37
Participants | 0

6. Secondary Outcome: 30-Day Post Operative Mortality
Description: The number of participants that died within 30 days of undergoing a pancreaticoduodenectomy.
Time Frame: 30 days after the time of surgery (Surgery is 28-42 days after start of treatment)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Beam Radiation/ Capecitabine
Number analyzed (Participants) | 37
Participants | 0

7. Secondary Outcome: Number of Participants With Treatment Related Serious Adverse Events
Description: The number of participants that had treatment related serious adverse events. Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE 3). Adverse events were considered to be serious adverse events if they were grade 3 or greater and were considered to be possibly, probably, or definitely related to treatment.
Time Frame: From the start of treatment until 30 days after the end of treatment, up to approximately 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Beam Radiation/ Capecitabine Dose Level 1 | Proton Beam Radiation/ Capecitabine Dose Level 2 | Proton Beam Radiation/ Capecitabine Dose Level 3 | Proton Beam Radiation/ Capecitabine Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 41
Participants | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment, up to approximately approximately 5 months
Arm/Group | Proton Beam Radiation/ Capecitabine Dose Level 1 | Proton Beam Radiation/ Capecitabine Dose Level 2 | Proton Beam Radiation/ Capecitabine Dose Level 3 | Proton Beam Radiation/ Capecitabine Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 2/41
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Beam Radiation/ Capecitabine Dose Level 1 (N=3) | Proton Beam Radiation/ Capecitabine Dose Level 2 (N=3) | Proton Beam Radiation/ Capecitabine Dose Level 3 (N=3) | Proton Beam Radiation/ Capecitabine Dose Level 4 (N=41)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Chest Wall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Beam Radiation/ Capecitabine Dose Level 1 (N=3) | Proton Beam Radiation/ Capecitabine Dose Level 2 (N=3) | Proton Beam Radiation/ Capecitabine Dose Level 3 (N=3) | Proton Beam Radiation/ Capecitabine Dose Level 4 (N=41)
Abdomen- pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (4) | 1 (4) | 9 (12)
ALT- SGPT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (3) | 2 (4) | 2 (4) | 7 (10)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
AST- SGOT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Back- pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Bilirubin (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (1) | 15 (23)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Fatigue (General disorders) | 3 (6) | 2 (4) | 3 (5) | 21 (33)
Fever w/o neutropenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (20)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4) | 3 (5) | 29 (43)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (2) | 7 (8)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-06-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT00438256/Prot_SAP_000.pdf